CLINICAL TRIAL: NCT03450109
Title: A Randomized and Open-label Study to Assess Pharmacokinetics, Pharmacodynamics and Safety of LY01005 Versus Goserelin Comparator (ZOLADEX®) Following a Single Administration in Patients With Prostate Cancer
Brief Title: A Study to Assess LY01005 Versus Goserelin Comparator (ZOLADEX®) in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LY01005/CT-USA-101
Record Dates: First submitted 2018-01-23; First posted 2018-03-01 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Cancer of Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LY01005 (Experimental): One LY01005 3.6 mg gluteal IM injection.
  Interventions: Drug: LY01005
- Zoladex (Active Comparator): One Zoladex 3.6 mg subcutaneous injection into the anterior abdominal wall
  Interventions: Drug: Zoladex

INTERVENTIONS:
Drug: LY01005 — One gluteal IM injection
  Arms: LY01005
Drug: Zoladex — One Subcutaneous injection in the abdominal wall
  Other Names: Goserelin
  Arms: Zoladex

SUMMARY:
A phase I, randomized, open-label and active-control study to assess the PK, PD and safety profiles of LY01005 versus goserelin comparator to be conducted in the USA.

DETAILED DESCRIPTION:
This will be a randomized, open-label and active-control study to assess the PK, PD and safety profiles of LY01005 versus goserelin comparator to be conducted in the USA.

ELIGIBILITY:
Inclusion Criteria:

1.Patient with an informed consent signed by the patient himself or legally acceptable representative before any trial-related activities; 2.2. Male patients diagnosed by confirmation of prostate cancer of any stages for whom endocrine treatment is indicated; patients with laboratory evidence of "biochemical recurrence" (BCR) are allowed. BCR is defined as the presence of prostate-specific antigen (PSA) greater than 0.2 ng/mL measured 6 to 13 weeks after radical prostatectomy followed by a confirmatory test showing persistent PSA greater than 0.2 ng/mL; or "PSA nadir + 2 ng/mL" (treated with radiation therapy); or PSA doubling time < 6 months without radiographic evidence of recurrence 3.Patients with a Screening testosterone level >1.5 ng/ml; 4.Patients with a life expectancy of at least 12 months; 5.Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2; 6.Patient understands and is willing to comply with the protocol and related procedures; 7.If having female sexual partners of childbearing potential, agree to avoid the occurrence of pregnancy during study participation and for 130 days after completing the study by using a highly effective method of contraception such as barrier method and female contraceptives, including spermicides, etc.

Exclusion Criteria:

1. Patients with a history of orchiectomy, adrenectomy or pituitary resection or receiving radiotherapy for prostate cancer (patients with prostatectomy are eligible for the study as are patients who received radiotherapy as long as radiotherapy was not received within 6 months prior to Screening);
2. Patients who have previously received hormonal therapy for prostate cancer, including surgical deprivation or sex hormone-regulating agents such as GnRH agonists/inhibitors as well as estrogen therapy. However, patients previously treated with neo-adjuvant therapy or adjuvant hormonal therapy for less than 6 months with an interval of at least 6 months since discontinuation of such therapy at the time of the Screening Visit can be enrolled;
3. Any patient at risk of urinary tract obstruction or spinal cord compression due to potential testosterone surge;
4. Patients with confirmed symptoms or signs related with to cerebral metastasis or radiographically confirmed brain metastases;
5. Patients with a history or presence of any other malignancy except recovered from basal cell carcinoma with no recurrence within the last 3 years;
6. Patients with a history of severe uncontrolled asthma, anaphylactic reactions, or severe urticaria and/or angioedema;
7. Patients with uncontrolled diabetes mellitus;
8. Patients with a history of hypersensitivity towards any components of the study drug;
9. Patients who test positive for drugs of abuse or alcohol, have smoked or otherwise used nicotine-containing products within 6 months prior to the Screening Visit, are smokers, drug abusers or have taken alcohol within 24 hours prior to dosing;
10. Patients who are taking medications for seizures or oral steroids such as dexamethasone, methylprednisolone or prednisone;
11. Patients who have taken 5α-reductase inhibitors (finasteride, dutasteride, and epristeride, etc.) within 3 months prior to Baseline Visit (Day 0);
12. Patients with an intellectual incapacity or language barrier precluding adequate understanding or co operation;
13. Patients who have received an investigational drug within the last 30 days before the Screening Visit or longer if considered to possibly influence the outcome of this trial;
14. Patients who are part of an ongoing trial;
15. Patients with an ECG at Screening of with a QTc >450 ms or have a family history of prolonged QT syndrome;
16. Patients with abnormal laboratory results which in the judgment of the investigator would affect the patient's health or the outcome of the trial;
17. Patients with a clinically significant medical condition (other than prostate cancer) including but not limited to: renal, hematological, gastrointestinal, endocrine, cardiac, neurological or psychiatric disease, alcohol or drug abuse or any other condition that may affect the patient's health or the outcome of the trial as judged by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
The bio-availability of goserelin in subjects receiving goserelin compared to Zoladex using Pharmacokinetic lab results | The pharmacokinetic (PK) labs will be drawn at -30 minutes of dosing, .25, .5, 1, and 6 hours of dosing and days 7, 10, 13, 16, 19, 22, 25, 29 and 36
  Area under the concentration-time curve (AUC) Assessment Area under the concentration-time curve (AUC) for the Pharmacokinetics (PK) of gosereling from LY01005 and goserelin from Zoladex will be determined.

SECONDARY OUTCOMES:
The bio-availability of goserelin in subjects receiving LY01005 compared to Zoladex using Pharmacodynamic lab results | The pharmacodynamic (PD) labs will be drawn at screening -30 minutes of dosing, .25, .5, 1, and 6 hours of dosing and days 2,4,7, 10, 13, 16, 19, 22, 25, 29 and 36
  Maximum concentration (Cmax) Assessment Maximum concentration (Cmax) for the Pharmacokinetics (PK) of goserelin from LY01005 and ODV from Zoladex will be determined.

OTHER OUTCOMES:
Safety profiles of LY01005 compared to goserelin comparator after a single injection | Safety parameters are collected at screening, days 0,2,4,7, 10, 13, 16, 19, 22, 25, 29,36, and follow up phone call
  Collection of adverse events throughout the study as a measure of safety and tolerability.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Pinnacle Research LLC, Anniston, Alabama
  - South Florida Medical Research, Aventura, Florida
  - Clinical Research Center of Flordia, Pompano Beach, Florida
  - Florida Urology Partners, Tampa, Florida
  - Urology, San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Zoladex Label — https://www.accessdata.fda.gov/drugsatfda_docs/label/2011/019726s054,020578s032lbl.pdf